CLINICAL TRIAL: NCT02202577
Title: Chlorhexidine-Alcohol Versus Povidone-Iodine for Surgical Site Antisepsis Prior to Cesarean Delivery
Brief Title: Chlorhexidine-Alcohol Versus Povidone-Iodine for Cesarean Antisepsis
Acronym: CAPICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPR-13-01063
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Surgical site antisepsis; Cesarean Delivery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ethanol; Paint; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine - Isopropyl alcohol (Experimental): Pre-operative skin preparation with Chlorhexidine Gluconate- Isopropyl alcohol
  Interventions: Drug: Chlorhexidine - Isopropyl alcohol
- Povidone-Iodine Scrub and Paint (Experimental): Pre-operative skin preparation with Povidone-Iodine Scrub and Paint
  Interventions: Drug: Povidone-Iodine Scrub and Paint

INTERVENTIONS:
Drug: Chlorhexidine - Isopropyl alcohol — Applied to skin pre-operatively for surgical site anti-sepsis; regulated as a drug by FDA
  Other Names: Chlora-Prep
  Arms: Chlorhexidine - Isopropyl alcohol
Drug: Povidone-Iodine Scrub and Paint — Applied to skin pre-operatively for surgical site anti-sepsis; regulated as a drug by FDA
  Other Names: Betadine
  Arms: Povidone-Iodine Scrub and Paint

SUMMARY:
Primary Hypothesis: chlorhexidine gluconate alcohol skin antiseptic preparation is superior to povidone-iodine scrub and paint skin antiseptic preparation for prevention of cesarean related surgical site infection.

DETAILED DESCRIPTION:
Patients who are considered likely to need cesarean delivery or who are planning cesarean will be recruited and consented for study participation during prenatal care and/or at time of admission to labor and delivery.

Patients undergoing cesarean who meet inclusion/exclusion criteria will be randomized to one of two surgical preparations as listed above (1. Chlorhexidine Gluconate (CHG)-alcohol, or 2. Povidone Iodine (P-I) scrub and paint. Randomization will be performed by the consenting surgeon (listed as key personnel) after the patient has arrived into the operating room for cesarean. Pre-operative surgical site antisepsis will be performed according to randomization. All other surgical practices will remain at the surgeon's discretion according to standard of care at Metrohealth.

Patients will be examined daily by the obstetric team and evaluated for signs and symptoms of surgical site infection, as standard in the investigators institution. The chart will be reviewed to determine if the patient was diagnosed during admission, or, re-admitted because of surgical site infection. The patient will also be questioned regarding any treatment or diagnosis of Surgical Site Infection (SSI) that occured after discharge to home at the routine six week post-operative visit. If patient does not return for the routine post-operative visit, the investigator will attempt to contact the patient by telephone to determine if the patient had been diagnosed or treated for surgical site infection. If patient is lost to 6 week follow up, subanalysis will be performed on available data derived from hospitalization and hospital Electronic Medical Record (EMR).

Data will be captured in RedCAP database.

Additional data will be captured that may affect patient likelihood of surgical site infection to ensure that both groups are statistically equal in risk factors for SSI: labor or rupture of membranes prior to cesarean, maternal age, estimated gestational age, Body Mass Index (BMI), gravity, parity, race, smoking status, hypertensive morbidity, diabetes, estimated blood loss, operative time, race, insurance type, general versus regional anesthesia, appropriate antibiotic prophylaxis given, skin closure (sutures v. staples).

Power analysis was performed: assuming 7.5% risk of cesarean site infection and a 50% reduction with chlorhexidine, 932 individuals will be recruited. Approximately 800 cesareans are performed at the investigators institution per year and the investigators anticipate that 80% will be eligible to participate.

Data review will be done every 6 months or every 200 patients and analyzed, whichever is sooner. Analysis will be performed by the Primary Investigators (PI) for completeness, accuracy, strict adherence to study protocol, safety, and statistical significance. The investigators site is also subject to periodic audits by the investigators Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* cesarean delivery
* age 18-65
* ability to consent in English or Spanish

Exclusion Criteria:

* inability or unwillingness to consent to study participation in English or Spanish
* current incarceration
* pre-operative diagnosis of chorioamnionitis
* perceived inability to complete follow up for data collection
* any prior known allergy or adverse reaction to either study preparation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian B Mercer, MD, Principal Investigator — MetroHealth Medical Center/Case Western Reserve; Edward H Springel, MD, Principal Investigator — MetroHealth Medical Center/Case Western Reserve
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252
- [Derived] Springel EH, Wang XY, Sarfoh VM, Stetzer BP, Weight SA, Mercer BM. A randomized open-label controlled trial of chlorhexidine-alcohol vs povidone-iodine for cesarean antisepsis: the CAPICA trial. Am J Obstet Gynecol. 2017 Oct;217(4):463.e1-463.e8. doi: 10.1016/j.ajog.2017.05.060. Epub 2017 Jun 7. PMID 28599898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and randomization began March 2014 and was successfully completed May 2016.
Period: Overall Study
Arm/Group | Chlorhexidine - Isopropyl Alcohol | Povidone-Iodine Scrub and Paint
Started | 461 | 471
Completed | 448 | 452
Not Completed | 13 | 19
Not completed — Lost to Follow-up | 6 | 16
Not completed — Protocol Violation | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine - Isopropyl Alcohol | Povidone-Iodine Scrub and Paint | Total
Number analyzed (Participants) | 461 | 471 | 932
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [24 to 33] | 28 [24 to 32] | 28 [24 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 471 | 932
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 207 | 210 | 417
  White | 182 | 186 | 368
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Surgical Site Infection
Description: Number of Patients with Cesarean-Related surgical site infection by Center for Disease Control (CDC) criteria: superficial, deep, organ space.
Time Frame: 4 weeks after cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine - Isopropyl Alcohol | Povidone-Iodine Scrub and Paint
Number analyzed (Participants) | 461 | 471
Participants | 29 | 33
Statistical Analysis 1: Comparison: Chlorhexidine - Isopropyl Alcohol vs Povidone-Iodine Scrub and Paint; We estimated a cesarean related surgical site infection rate of 7.5% with povidone-iodine and hypothesized chlorhexidine-alcohol treatment to be superior based on existing literature. We considered a 50% reduction to be significant. We performed our power analysis assuming 1-directional effects in favor of chlorhexidine, which best fit our hypothesis. Using a 1-tailed alpha of 0.05 and an 80% power to detect a difference, we estimated that 466 subjects would be required in each group; Test type: Superiority; p = 0.38, Fisher Exact — This is the calculated p-value for the intention to treat analysis of primary outcome. A 1-tailed p value of <0.05 was selected for statistical significance; Risk Ratio (RR) = 0.90, 95% CI 1-sided [upper limit 1.35]
Statistical Analysis 2: Comparison: Chlorhexidine - Isopropyl Alcohol vs Povidone-Iodine Scrub and Paint; Per Protocol Analysis; Test type: Superiority; p = 0.26, Fisher Exact — This is the calculated p-value for the per protocol analysis of primary outcome. A 1-tailed p value of <0.05 was selected for statistical significance; Risk Ratio (RR) = 0.83, 95% CI 1-sided [upper limit 1.25]

2. Secondary Outcome: Number of Patients With Non-infections Surgical Site Complications
Description: Non-infection complications: allergic skin reactions, hematomas, wound separation, dehiscence.
Time Frame: 4 weeks after cesarean delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine - Isopropyl Alcohol | Povidone-Iodine Scrub and Paint
Number analyzed (Participants) | 461 | 471
Participants | 19 | 17

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse event data was collected at the same time as primary outcome data.
Arm/Group | Chlorhexidine - Isopropyl Alcohol | Povidone-Iodine Scrub and Paint
All-Cause Mortality (participants affected / at risk) | 0/461 | 0/471
Serious Adverse Events (participants affected / at risk) | 0/461 | 0/471
Other Adverse Events (participants affected / at risk) | 0/461 | 0/471

LIMITATIONS AND CAVEATS:
Lack of masking of clinical personnel to treatment assignment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No